CLINICAL TRIAL: NCT01906658
Title: A Study to Explore the Safety and Tolerability of Acthar in Patients With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QSC01-ALS-01
Record Dates: First submitted 2013-07-15; First posted 2013-07-24 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: H.P. Acthar Gel; Acthar; amyotrophic lateral sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acthar 80 U (1.0 mL) SC twice weekly (Experimental): Acthar (Repository Corticotropin Injection) 80 U (1.0 mL) SC twice weekly
  Interventions: Drug: Repository corticotropin injection
- Acthar 24 U (0.3 mL) SC daily (Experimental): Acthar (Repository Corticotropin Injection) 24 U (0.3 mL) SC daily
  Interventions: Drug: Repository corticotropin injection
- Acthar 56 U (0.7 mL) SC twice weekly (Experimental): Acthar (Repository Corticotropin Injection) 56 U (0.7 mL) SC twice weekly
  Interventions: Drug: Repository corticotropin injection
- Acthar 16 U (0.2 mL) SC daily (Experimental): Acthar (Repository Corticotropin Injection) 16 U (0.2 mL) SC daily
  Interventions: Drug: Repository corticotropin injection

INTERVENTIONS:
Drug: Repository corticotropin injection — Acthar given SC twice weekly (80 U or 56 U) or daily (24 U or 16 U) for 8 weeks
  Other Names: H.P. Acthar Gel; Acthar; ACTH Gel; ACTH

SUMMARY:
This 8-week randomized, open-label evaluation will examine the acute safety and tolerability of 4 different dosing regimens of Acthar to inform dose selection for future studies of Acthar in patients with Amyotrophic Lateral Sclerosis (ALS). The study will also investigate the mean rate of change in the ALSFRS-R total score as an exploratory endpoint to help design future studies.

This study will enroll up to 40 patients and include an optional 28-week open-label extension period plus a 3-week treatment taper and 1-week follow up period. After completion of Week 8, patients enrolled in a treatment group that is considered safe and tolerable at that time have the option to continue into the open-label extension period. A 3-week treatment taper and a follow-up visit are planned for all patients enrolled in the study, beginning either at Week 8 or at Week 36 if a patient continues into the optional open-label extension period.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Diagnosis of clinically definite ALS, clinically probable-laboratory supported ALS, clinically probable ALS, or clinically possible ALS based on the revised El Escorial criteria.
* Patients with ALS ≤ 3 years since symptom onset. Symptom onset is defined as date of first muscle weakness or dysarthria.
* Upright slow vital capacity (SVC)≥ 60% of predicted.
* If taking riluzole and/or Nuedexta®, stable regimen is required for ≥ 30 days prior to screening.
* Medically (either independently or with caregiver assistance) able to comply with study procedures, including subcutaneous (SC) injections of study medication and adherence to concomitant medication restrictions.

Exclusion Criteria:

* Any medical condition known to have an association with motor neuron dysfunction which might confound or obscure the diagnosis of ALS.
* Tracheostomy, diaphragm pacing, or ongoing need for assisted ventilation of any type (e.g., bilevel positive airway pressure) for treatment of ALS-related respiratory dysfunction (vital capacity of < 60% predicted, nocturnal desaturation, and/or nocturnal hypoventilation). Patients on assisted ventilation for other reasons require approval from the Medical Monitor. (Supplemental oxygen is acceptable).
* Recorded diagnosis or evidence of major psychiatric disorder.
* Clinically evident cognitive and/or behavioral impairment that in the opinion of the Investigator would impair the ability of the patient to comply with the study procedures.
* Therapies and/or Medications:

  1. History of prior sensitivity to Acthar or other porcine protein products.
  2. Chronic systemic corticosteroid use, defined as > 20 mg of prednisone or equivalent systemic corticosteroid taken for more than 4 consecutive weeks within 6 months prior to randomization. Topical, inhaled, or intra-articular corticosteroids are allowed.
  3. Planned treatment with live or live attenuated vaccines once enrolled in the study.
* Participation in another therapeutic (drug or device) investigational study within 30 days prior to screening.
* Type 1 or type 2 diabetes mellitus, or patients currently taking hypoglycemic medication.
* Contraindication per Acthar Prescribing Information, Appendix D Section 4: scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of peptic ulcer, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency, or adrenal cortical hyperfunction.

  1. For the purposes of this study, osteoporosis is defined as a history of a lumbar spine and/or femoral neck T-score ≤ -2.5 on bone densitometry (DXA), OR osteoporosis requiring pharmacologic therapy, OR a history of non-traumatic low impact hip or vertebral fracture, OR patient reported history of osteoporosis.
  2. For the purposes of this study, history of peptic ulcer is defined as ≤ 6 months prior to screening.
  3. For the purposes of this study, uncontrolled hypertension is defined as mean systolic blood pressure ≥ 140 mmHg and diastolic blood pressure ≥ 90 mmHg on ≥ 3 seated readings taken at least 5 minutes apart during the screening period.
  4. For the purposes of this study, congestive heart failure is defined as New York Heart Association Functional Class III-IV.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Questcor Investigational Site, Birmingham, Alabama
  - Questcor Investigational Site, Phoenix, Arizona
  - Questcor Investigational Site, San Francisco, California
  - Questcor Investigational Site, Stanford, California
  - Questcor Investigational Site, Jacksonville, Florida
  - Questcor Investigational Site, Miami, Florida
  - Questcor Investigational Site, Tampa, Florida
  - Questcor Investigational Site, Atlanta, Georgia
  - Questcor Investigational Site, Kansas City, Kansas
  - Questcor Investigational Site, Rochester, Minnesota
  - Questcor Investigational Site, Lincoln, Nebraska
  - Questcor Investigational Site, Hershey, Pennsylvania
  - Questcor Investigational Site, Pittsburgh, Pennsylvania
  - Questcor Investigational Site, Memphis, Tennessee
  - Questcor Investigational Site, Dallas, Texas
  - Questcor Investigational Site, Houston, Texas
  - Questcor Investigational Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Acthar 80 U (1.0 mL) Subcutaneous (SC) Twice Weekly: Acthar (Repository Corticotropin Injection) 80 U (1.0 mL) SC twice weekly
  Repository corticotropin injection: Acthar given SC twice weekly (80 U or 56 U) or daily (24 U or 16 U) for 8 weeks
Period: Overall Study
Arm/Group | Acthar 80 U (1.0 mL) Subcutaneous (SC) Twice Weekly | Acthar 24 U (0.3 mL) SC Daily | Acthar 56 U (0.7 mL) SC Twice Weekly | Acthar 16 U (0.2 mL) SC Daily
Started | 11 | 11 | 10 | 11
Completed | 9 | 10 | 7 | 11
Not Completed | 2 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acthar 80 U (1.0 mL) SC Twice Weekly | Acthar 24 U (0.3 mL) SC Daily | Acthar 56 U (0.7 mL) SC Twice Weekly | Acthar 16 U (0.2 mL) SC Daily | Total
Number analyzed (Participants) | 11 | 11 | 10 | 11 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 6 | 9 | 26
  >=65 years | 7 | 4 | 4 | 2 | 17
Gender [Count of Participants; unit: Participants]
  Female | 4 | 5 | 4 | 4 | 17
  Male | 7 | 6 | 6 | 7 | 26
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 10 | 11 | 43

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Adverse Events (AEs) That Required Study Drug Discontinuation or Could Not be Controlled With Concomitant Medication
Time Frame: Baseline to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar 80 U (1.0 mL) SC Twice Weekly | Acthar 24 U (0.3 mL) SC Daily | Acthar 56 U (0.7 mL) SC Twice Weekly | Acthar 16 U (0.2 mL) SC Daily
Number analyzed (Participants) | 11 | 11 | 10 | 11
Participants | 2 | 0 | 2 | 0

2. Secondary Outcome: Proportion of Subjects With Adverse Events That Required Study Drug Discontinuation
Time Frame: Baseline to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar 80 U (1.0 mL) SC Twice Weekly | Acthar 24 U (0.3 mL) SC Daily | Acthar 56 U (0.7 mL) SC Twice Weekly | Acthar 16 U (0.2 mL) SC Daily
Number analyzed (Participants) | 11 | 11 | 10 | 11
Participants | 2 | 0 | 2 | 0

3. Secondary Outcome: Proportion of Subjects With Adverse Events That Could Not be Controlled by Concomitant Medication
Time Frame: Baseline to Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar 80 U (1.0 mL) SC Twice Weekly | Acthar 24 U (0.3 mL) SC Daily | Acthar 56 U (0.7 mL) SC Twice Weekly | Acthar 16 U (0.2 mL) SC Daily
Number analyzed (Participants) | 11 | 11 | 10 | 11
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Proportion of Subjects With Treatment Emergent Suicidality
Time Frame: Baseline to Week 36
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar 80 U (1.0 mL) SC Twice Weekly | Acthar 24 U (0.3 mL) SC Daily | Acthar 56 U (0.7 mL) SC Twice Weekly | Acthar 16 U (0.2 mL) SC Daily
Number analyzed (Participants) | 11 | 11 | 10 | 11
Participants | 1 | 3 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Acthar 80 U (1.0 mL) SC Twice Weekly | Acthar 24 U (0.3 mL) SC Daily | Acthar 56 U (0.7 mL) SC Twice Weekly | Acthar 16 U (0.2 mL) SC Daily
Serious Adverse Events (participants affected / at risk) | 2/11 | 3/11 | 1/10 | 1/11
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11 | 9/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acthar 80 U (1.0 mL) SC Twice Weekly (N=11) | Acthar 24 U (0.3 mL) SC Daily (N=11) | Acthar 56 U (0.7 mL) SC Twice Weekly (N=10) | Acthar 16 U (0.2 mL) SC Daily (N=11)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acthar 80 U (1.0 mL) SC Twice Weekly (N=11) | Acthar 24 U (0.3 mL) SC Daily (N=11) | Acthar 56 U (0.7 mL) SC Twice Weekly (N=10) | Acthar 16 U (0.2 mL) SC Daily (N=11)
Edema, peripheral (General disorders) | 4 | 2 | 2 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5 | 4
Headache (Nervous system disorders) | 0 | 3 | 5 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 5
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 2 | 2
Asthenia (General disorders) | 4 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 3
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 1 | 3 | 2
Anxiety (Psychiatric disorders) | 3 | 0 | 2 | 1
Edema (General disorders) | 2 | 3 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 3
Vision blurred (Eye disorders) | 1 | 2 | 0 | 3
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator shall not, without Sponsor's prior written consent, independently publish or otherwise disclose any results of the study until a Multi-Center Publication is published. If a Multi-Center Publication is not submitted for publication within the specified timeframe, Institution and Principal Investigator shall have the right to publish and present the results of Institution's and Principal Investigator's activities solely in accordance with the Sponsor's written provisions.